CLINICAL TRIAL: NCT00653913
Title: Evaluation of Potential for Pharmacokinetic Drug Interaction Between SCH 58235 and Pitavastatin
Brief Title: Evaluation of Potential for Drug Interaction Between SCH 58235 (Ezetimibe) and Pitavastatin (Study P03962)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P03962
Record Dates: First submitted 2008-03-31; First posted 2008-04-07 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A (Active Comparator): SCH 58235 (Period 1) Pitavastatin (Period 2) Coadministration (Period 3)
  Interventions: Drug: SCH 58235; Drug: pitavastatin
- Group B (Active Comparator): SCH 58235 (Period 1) Coadministration (Period 2) Pitavastatin (Period 3)
  Interventions: Drug: SCH 58235; Drug: pitavastatin
- Group C (Active Comparator): Pitavastatin (Period 1) SCH 58235 (Period 2) Coadministration (Period 3)
  Interventions: Drug: SCH 58235; Drug: pitavastatin
- Group D (Active Comparator): Pitavastatin (Period 1) Coadministration (Period 2) SCH 58235 (Period 3)
  Interventions: Drug: SCH 58235; Drug: pitavastatin
- Group E (Active Comparator): Coadministration (Period 1) SCH 58235 (Period 2) Pitavastatin (Period 3)
  Interventions: Drug: SCH 58235; Drug: pitavastatin
- Group F (Active Comparator): Coadministration (Period 1) Pitavastatin (Period 2) SCH 58235 (Period 3)
  Interventions: Drug: SCH 58235; Drug: pitavastatin

INTERVENTIONS:
Drug: SCH 58235 — SCH 58235 10 mg (once daily)
  Other Names: Ezetimibe
Drug: pitavastatin — Pitavastatin 2 mg (once daily)

SUMMARY:
This study was designed to evaluate the pharmacokinetic interaction and safety of coadministration of SCH 58235 (ezetimibe) and pitavastatin in healthy Japanese adult male subjects or adult male subjects having no obvious disease other than high cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects meeting all the criteria below or adult male subjects having no obvious disease other than high cholesterol levels.
* Aged 20 years or over and 65 years or below when the informed consent is obtained.
* Weighing 50 kg or over and 80 kg or below on the day of the screening tests, with BMI [Body Mass Index: body weight (kg)/height (m)2] ranging from 16.5 to 27.5.

Exclusion Criteria:

Patients meeting any one of the following conditions are excluded from the study.

* Subjects with the triglyceride value at screening test exceeding 500 mg/dL.
* Subjects with past history of drug allergy (shock, anaphylactic symptom, and angioedema).
* Subjects with past history of alcohol or drug dependence.
* Subjects with past history of mental disorder.
* Subjects positive in the test for HBs antigen, HCV antibody, or HIV antibody or in the serological test for syphilis.
* Subjects who used any drug within 2 weeks of investigational product administration in Period 1.
* Subjects who have drawn more than 400 mL of blood within 12 weeks before administration day in Period 1.
* Subjects who participated in other study within 16 weeks of investigational product administration in Period 1 and was administered a investigational product.
* Subjects who cannot take contraceptive measures during the study period (from providing informed consent to completion of Period 3 examination)
* Subjects who the investigator judges are inappropriate to participate in the study.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-03; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Compare plasma concentrations of SCH 58235 (ezetimibe) and pitavastatin after administration of each drug alone and in combination, using Cmax and AUC(0-24h). | Day 7 of each period

SECONDARY OUTCOMES:
Compare plasma concentrations of SCH 58235 (ezetimibe) and pitavastatin administration of each drug alone and in coadministration, using Tmax, plasma concentration 24 h after last dose, and AUC(I). | Day 7 of each period
Adverse events, laboratory tests results, and vital signs. | Throughout study